CLINICAL TRIAL: NCT02090153
Title: Phase II Study of S-1 Plus Leucovorin (1 Week on and 1 Week Off) as First-line Treatment for Patients With Metastatic and Recurrent Gastric Cancer
Brief Title: Study of S-1 Plus LV for Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ruihua Xu, vice president of SunYat-sen University Cancer Center,head of medical oncology department, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL for AGC
Record Dates: First submitted 2014-03-12; First posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Gastric Cancer
Keywords: Advance Gastric Cancer,; S-1 plus leucovorin,; ORR,; OS,; TTP,; TTF,; Adverse events,; Pharmacokinetics
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Tegafur; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S-1 plus LV (Experimental): All patients were orally treated with S-1 in doses of 40 mg (body surface area (BSA)<1.25 m2), 50 mg (1.25≤BSA<1.50 m2) and 60 mg (BSA≥1.50 m2) b.i.d. on days 1-7 in combination with LV given simultaneously at a ﬁxed dose of 25 mg b.i.d. on days 1-7, followed by a 7 day rest. Treatment courses were repeated every 2 weeks.
  Interventions: Drug: S-1; Drug: LV

INTERVENTIONS:
Drug: S-1 — 40~60mg bid，d1~7 q2W
  Other Names: tegafur/gimeracil/oteracil potassium
Drug: LV — LV is given simultaneously at a ﬁxed dose of 25 mg b.i.d. on days 1-7, followed by a 7 day rest.
  Other Names: Leucovorin

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of S-1 plus Leucovorin (1 week on and 1 week off) as first-line treatment for patients with metastatic and recurrent gastric cancer.

DETAILED DESCRIPTION:
Patients enrolled in this study were orally treated with S-1 in doses of 40 mg (body surface area (BSA)<1.25 m2), 50 mg (1.25≤BSA<1.50 m2) and 60 mg (BSA≥1.50 m2) b.i.d. on days 1-7 in combination with LV given simultaneously at a ﬁxed dose of 25 mg b.i.d. on days 1-7, followed by a 7 day rest. Treatment courses were repeated every 2 weeks. Treatment was continued until progressive disease (PD), unacceptable toxicity or patient refusal.

ELIGIBILITY:
Inclusion Criteria:

* histologically conﬁrmed metastatic or recurrent gastric cancer
* with at least one measurable lesion by RECIST criteria
* an age of ≥ 18
* adequate oral intake
* no previous radiotherapy, immunotherapy, biotherapy, hormonotherapy and chemotherapy within 5 years (adjuvant chemotherapy without S-1 was allowed if ﬁnished 6 months before enrollment)
* an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* adequate bone marrow function, hepatic function and renal functions

Exclusion Criteria:

* a history of hypersensitivity to S-1 or LV, usage of drugs interacting with S-1
* serious concomitant conditions (severe heart disease, pulmonary ﬁbrosis, intestinal obstruction, enteroplegia, renal failure, liver failure, pre-existing sensory neuropathy ≥ grade 2, uncontrolled infections, psychogenic disorders, human immunodeﬁciency virus infection, severe diarrhea, nausea, or vomiting, severe ascites or pleural effusion, etc.)
* extensive bone metastasis, brain metastasis or meningeal metastasis
* another synchronous cancer
* surgery within 3 weeks before enrollment
* participating in other clinical studies
* women who were or to be pregnant, nursing infants, and men who were to conceive children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 1 year
  The primary endpoint is overall response rate,which equals the rate of patients with CR+PR.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 1-1.5 years
  Progression-free survival (PFS) was determined from the date of treatment to progression or death
Overall survival (OS) | 1-2.5 years
  Overall survival (OS) was calculated from the date of treatment to death from any cause or the last date of follow-up.
Time to treatment failure (TTF) | 1 year
  Time to treatment failure (TTF) was determined from the date of treatment to progression, death, refusal or interruption due to adverse events.
Disease control rate | 1 year
  Disease control rate equals the rate of patients with CR+PR+SD.
Adverse Events (AEs) | 2 year
  All treatment-related adverse events (AEs) were categorized according to the National Cancer Institute's Common Terminology Criteria for Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Professor, Principal Investigator — SunYat-sen University Cancer Center
Locations (1):
- Sun Yat-sen University Cancer Center, Gaungzhou, Guangdong, China

REFERENCES:
- [Background] Koizumi W, Boku N, Yamaguchi K, Miyata Y, Sawaki A, Kato T, Toh Y, Hyodo I, Nishina T, Furuhata T, Miyashita K, Okada Y. Phase II study of S-1 plus leucovorin in patients with metastatic colorectal cancer. Ann Oncol. 2010 Apr;21(4):766-771. doi: 10.1093/annonc/mdp371. Epub 2009 Oct 14. PMID 19828562
- [Derived] He MM, Zhang DS, Wang F, Wang ZX, Yuan SQ, Wang ZQ, Luo HY, Ren C, Qiu MZ, Jin Y, Wang DS, Chen DL, Zeng ZL, Li YH, He YY, Hao YT, Guo P, Wang FH, Zeng YX, Xu RH. Phase II trial of S-1 plus leucovorin in patients with advanced gastric cancer and clinical prediction by S-1 pharmacogenetic pathway. Cancer Chemother Pharmacol. 2017 Jan;79(1):69-79. doi: 10.1007/s00280-016-3209-1. Epub 2016 Dec 2. PMID 27913881
- See also: Long-term outcomes and prognostic factors of patients with advanced gastric cancer treated with S-1 plus cisplatin combination chemotherapy as a first-line treatment. — http://www.ncbi.nlm.nih.gov/pubmed/23999902
- See also: S-1-Based Chemotherapy versus Capecitabine-Based Chemotherapy as First-Line Treatment for Advanced Gastric Carcinoma: A Meta-Analysis. — http://www.ncbi.nlm.nih.gov/pubmed/24349363